CLINICAL TRIAL: NCT00036218
Title: A Phase III, Double-Blind, Placebo-Controlled, Randomized Study Comparing the Efficacy, Safety, and Tolerability of Sumanirole Versus Placebo or Ropinirole in Patients With Early Parkinson's Disease.
Brief Title: Study Evaluating Sumanirole for the Treatment of the Signs and Symptoms of Early Parkinson's Disease.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 666E-CNS-0075-021
Record Dates: First submitted 2002-05-08; First posted 2002-05-09 (Estimated); Last update posted 2006-06-07 (Estimated); Status verified 2006-06

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease | interventions — U 95666E; ropinirole

INTERVENTIONS:
Drug: sumanirole
Drug: ropinirole

SUMMARY:
The primary purpose of this study is to determine whether sumanirole is effective and safe in the treatment of the signs and symptoms of early Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

Parkinson's disease of less than 7 years duration

Modified Hoehn and Yahr Scale Stages 1 through 3.

Age greater than or equal to 30 years old.

Men or women (women of childbearing potential must have a negative pregnancy test at screen) and both must use adequate contraceptive methods.

Patients who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.

Exclusion Criteria:

Atypical Parkinson's disease syndromes due to drugs, metabolic disorders, encephalitis, or degenerative diseases.

Levodopa received for 1-year accumulated interval in the last two years.

Dopamine agonist medications or catechol-o-methyl transferase inhibitors in the 30 days prior to baseline.

Unstable dose regimes of hypnotics, anxiolytics or antidepressants

Dementia

History of stereotaxic brain surgery, psychosis or active epilepsy within past year.

Participation in clinical trial within the previous 30 days.

Malignant melanoma or history of melanoma

Significant medical or pshychiatric condition.

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600
Dates: Start 2001-12; Study Completion 2003-04

PRIMARY OUTCOMES:
Change from baseline in UPDRS (Unified Parkinson's Disease Rating Scale) II + III total scores at end of maintenance, for sumanirole compared to placebo

SECONDARY OUTCOMES:
To assess the safety profile of sumanirole; the benefit of sumanirole in quality of life measures, and change from baseline in UPDRS II + III total scores at end of maintenance, for sumanirole compared to ropinirole

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (90):
- United States (84):
  - Pfizer Investigational Site, Hot Springs, Arkansas
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Carmichael, California
  - Pfizer Investigational Site, Fresno, California
  - Pfizer Investigational Site, Irvine, California
  - Pfizer Investigational Site, La Jolla, California
  - Pfizer Investigational Site, Loma Linda, California
  - Pfizer Investigational Site, Los Angeles, California
  - Pfizer Investigational Site, Oceanside, California
  - Pfizer Investigational Site, San Francisco, California
  - Pfizer Investigational Site, San Luis Obiapo, California
  - Pfizer Investigational Site, Walnut Creek, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Fairfield, Connecticut
  - Pfizer Investigational Site, New Haven, Connecticut
  - Pfizer Investigational Site, Wilmington, Delaware
  - Pfizer Investigational Site, Boca Raton, Florida
  - Pfizer Investigational Site, Clearwater, Florida
  - Pfizer Investigational Site, Fort Lauderdale, Florida
  - Pfizer Investigational Site, Jacksonville, Florida
  - Pfizer Investigational Site, Maitland, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Orlando, Florida
  - Pfizer Investigational Site, Palm Beach Gardens, Florida
  - Pfizer Investigational Site, Plantation, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Tampa, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Conyers, Georgia
  - Pfizer Investigational Site, Decatur, Georgia
  - Pfizer Investigational Site, Savannah, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Glenbrook, Illinois
  - Pfizer Investigational Site, Kansas City, Kansas
  - Pfizer Investigational Site, Lake Charles, Louisiana
  - Pfizer Investigational Site, Shreveport, Louisiana
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Columbia, Maryland
  - Pfizer Investigational Site, Frederick, Maryland
  - Pfizer Investigational Site, Rockville, Maryland
  - Pfizer Investigational Site, Boston, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, East Lansing, Michigan
  - Pfizer Investigational Site, Grand Rapids, Michigan
  - Pfizer Investigational Site, Southfield, Michigan
  - Pfizer Investigational Site, Traverse City, Michigan
  - Pfizer Investigational Site, Golden Valley, Minnesota
  - Pfizer Investigational Site, Minneapolis, Minnesota
  - Pfizer Investigational Site, Saint Cloud, Minnesota
  - Pfizer Investigational Site, Kansas City, Missouri
  - Pfizer Investigational Site, Springfield, Missouri
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Henderson, Nevada
  - Pfizer Investigational Site, Lebanon, New Hampshire
  - Pfizer Investigational Site, Morristown, New Jersey
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Ridgewood, New Jersey
  - Pfizer Investigational Site, Manhasset, New York
  - Pfizer Investigational Site, Mineola, New York
  - Pfizer Investigational Site, Mount Vernon, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Asheville, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Norristown, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, Upland, Pennsylvania
  - Pfizer Investigational Site, Knoxville, Tennessee
  - Pfizer Investigational Site, Memphis, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Salt Lake City, Utah
  - Pfizer Investigational Site, Burlington, Vermont
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Bellevue, Washington
  - Pfizer Investigational Site, Spokane, Washington
  - Pfizer Investigational Site, Wenatchee, Washington
  - Pfizer Investigational Site, Milwaukee, Wisconsin
- Argentina (3):
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires
  - Pfizer Investigational Site, Mar del Plata, Buenos Aires
  - Pfizer Investigational Site, Buenos Aires, Buenos Aires F.D.
- Mexico (2):
  - Pfizer Investigational Site, Mexico City, Mexico City
  - Pfizer Investigational Site, Monterrey, Nuevo León
- Pfizer Investigational Site, Carolina, Puerto Rico

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=666E-CNS-0075-021&StudyName=Study+evaluating+sumanirole+for+the+treatment+of+the+signs+and+symptoms+of+early+Parkinson%27s+disease%2E